CLINICAL TRIAL: NCT06032494
Title: Neo-vital: Investigating Changes in Vital Signs in Neonates
Brief Title: Investigating Changes in Vital Signs in Neonates
Acronym: Neo-vital
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: PID16761
Record Dates: First submitted 2023-08-09; First posted 2023-09-13 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Infant; Newborn
Keywords: preterm; respiration; oxygen saturation; heart rate
MeSH Terms: conditions — Premature Birth; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1 in 7 babies require neonatal care. During their time in hospital their vital signs (such as heart rate, breathing rate and oxygen saturation) are continuously monitored as part of standard care. Many factors lead to changes in vital signs, for example, medical procedures such as blood tests can result in brief increases in heart rate. Medication can also alter vital signs, either as an intended effect or as a side effect. However, different infants will respond in different ways to both procedures and medication. Predicting how an individual infant may respond could lead to better individualised care for infants. For example, using an infant's baseline vital signs to predict whether they will experience cardiorespiratory side effects from a particular drug could mean that doctors could choose an alternative safer treatment plan. To develop these predictive models, it is essential to first better understand how infants' vital signs are affected by different procedures and drugs, and how these effects are impacted by other factors such as infection, other pathologies, interaction between drugs and age.

Despite their routine use in hospital neonatal units, detailed electronic records of vital signs are often not recorded. Often, only major events or average values are stated on clinical records. Subtle changes in vital signs are therefore missed, and more complex analysis that may reveal important predictive features within the data is not possible. In this study the investigators will electronically record infant vital signs across longer time periods and during a variety of clinically-necessary procedures and administration of drugs, to explore how these impact vital signs and are altered by factors such as age and pathology. These will be compared with control procedures, such as a nappy change, or when the infant is resting in their cot or receiving skin-to-skin care.

ELIGIBILITY:
Inclusion Criteria:

Infants will be eligible to be included in the study if they are:

* Born to, or expected to be born to, a mother aged 16 or over
* Admitted to the Newborn Care Unit, John Radcliffe Hospital, or anticipated delivery of a baby who will require admittance to the Newborn Care Unit at birth
* Mother given informed written consent

Exclusion Criteria:

Infants will be ineligible if the following exclusion criteria applies:

• Known chromosomal abnormality or life-threatening congenital abnormality

Max Age: 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This single-centre prospective observational exploratory study will take place at the John Radcliffe Hospital, Oxford. Participants will be infants receiving inpatient care on the Newborn Care Unit.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in heart rate following drug administration | 1 day after drug administration, compared with baseline of 1 day before drug administration.
  To characterise the change in heart rate in infants following drug administration in a wide range of commonly used drugs in neonatal care. Drugs will only be administered as part of clinical care, no drugs are administered for research purposes
Change in oxygen saturation following drug administration | 1 day after drug administration, compared with baseline of 1 day before drug administration.
  To characterise the change in oxygen saturation in infants following drug administration in a wide range of commonly used drugs in neonatal care. Drugs will only be administered as part of clinical care, no drugs are administered for research purposes
Change in respiratory rate following drug administration | 1 day after drug administration, compared with baseline of 1 day before drug administration.
  To characterise the change in heart rate in infants following drug administration in a wide range of commonly used drugs in neonatal care. Drugs will only be administered as part of clinical care, no drugs are administered for research purposes
Change in heart rate following procedures | 1 day after procedure, compared with baseline of 1 day before procedure.
  To characterise the change in heart rate in infants in relation to procedures, including (but not limited to) intubation and extubation, LISA (less invasive surfactant administration), blood transfusion and acute medically-required painful procedures.
Change in oxygen saturation following procedures | 1 day after procedure, compared with baseline of 1 day before procedure.
  To characterise the change in oxygen saturation in infants in relation to procedures, including (but not limited to) intubation and extubation, LISA (less invasive surfactant administration), blood transfusion and acute medically-required painful procedures.
Change in respiratory rate following procedures | 1 day after procedure, compared with baseline of 1 day before procedure.
  To characterise the change in respiratory rate in infants in relation to procedures, including (but not limited to) intubation and extubation, LISA (less invasive surfactant administration), blood transfusion and acute medically-required painful procedures.

SECONDARY OUTCOMES:
Models of drug response | 1 day after drug administration, compared with baseline of 1 day before drug administration.
  Prediction of drug regimen requirements in individual infants from respiratory rate.
Models of procedure response | 1 day after procedure, compared with baseline of 1 day before procedure.
  Prediction of procedure outcome in individual infants (e.g. extubation success) from respiratory rate

CONTACTS AND LOCATIONS:
Locations (1):
- John Radcliffe Hospital, Oxford, United Kingdom